CLINICAL TRIAL: NCT02461407
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Clinical Trial to Compare the Efficacy and Safety of Anlotinib Versus Placebo in Patients With Gastric Cancer(ALTER0503)
Brief Title: Study of Anlotinib in Patients With Gastric Cancer(ALTER0503)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALTN-05-II
Record Dates: First submitted 2015-06-01; First posted 2015-06-03 (Estimated); Last update posted 2017-12-29 (Actual); Status verified 2017-08

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Anlotinib (Experimental): Anlotinib QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Anlotinib
- Placebo (Placebo Comparator): Placebo QD po and it should be continued until disease progression or intolerable toxicity or patients withdrawal of consent
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Anlotinib p.o. qd
  Arms: Anlotinib
Drug: Placebo — Placebo p.o. qd
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the effects and safety of Anlotinib with placebo in patients with Gastric Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent;
2. Pathologically confirmed advanced gastric adenocarcinoma (including Gastroesophageal junction adenocarcinoma) with measurable lesions outside stomach (RECIST 1.1)
3. Advanced stomach cancer patients who have failed to the second line or higher line chemotherapy treatment
4. >=18 years old；ECOG PS：0~1；Estimated life expectancy >3 months
5. Main organs function is normal;

Exclusion Criteria:

1. Patients who have been treated with anlotinib previously;
2. Patients who have been treated with other VEGFR-TKI small-molecule drugs previously, such as sunitinib, Sorafenib, famitinib, Apatinib, Regorafenib, ect
3. Patients suffering from other malignancies currently or within 5 years, except for cured cervical carcinoma in situ, non-melanoma skin cancers and superficial bladder cancer [ Ta (non-invasive carcinoma), Tis (carcinoma in situ) and T1 (carcinoma invasion into lamina propria) ]
4. Systemic anti-cancer therapy scheduled 4 weeks prior to assignment or during this study，including cytotoxic therapy，signal transduction inhibitors，immunotherapy(or received mitomycin C within 6 weeks before this study). Extended field radiotherapy(EF-RT) used within 4 weeks prior to assignment or limited field radiotherapy used to assess tumor lesions within 2 weeks prior to assignment;
5. CTCAE(4.0) Grade 1 or higher non-remission toxicity induced by any other previous treatments，excluding alopecia and Grade 2 or lower neurotoxicity induced by oxaliplatin;
6. Patients with a clear tendency of gastrointestinal bleeding;
7. Patients with factors that could affect oral medication (such as dysphagia，chronic diarrhea etc.)
8. Patients with pleural effusion or ascites, causing respiratory syndrome (CTCAE Grade 2 or higher dyspnea [Grade 2 dyspnea refers to Shortness of breath with a small amount of activities, affecting Instrumental activities of daily life])
9. Patients with any severe and/or unable to control diseases;
10. Patients underwent major surgical treatment，open biopsy or significant traumatic injury within 28 days prior to assignment;
11. Patients with any physical signs of bleeding diathesis or medical history, no matter how serious degree they are; Patients with any CTCAE Grade 3 or higher bleeding events occurred within 4 weeks prior to assignment; Patients with non-healing wounds，ulcers or fractures;
12. Patients with arterial or venous thromboembolic events occurred within 6 months, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis and pulmonary embolism;
13. Patients with drug abuse history and unable to get rid of or Patients with mental disorders
14. Brain metastases patients with symptoms or symptoms controlled < 2 months;
15. Patients participated in other anticancer drug clinical trials within 4 weeks or Patients participating in other clinical trials now;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2015-06 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From randomization until death (up to 24 months)

SECONDARY OUTCOMES:
Progress free survival (PFS) | each 42 days up to PD or death(up to 24 months)
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)

CONTACTS AND LOCATIONS:
Locations (38):
- China (38):
  - The First Affiliated Hospital, Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The 307th Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - Chongqing Daping Hospital, Chongqing, Chongqing Municipality
  - Union Hospital of Fujian Medical University, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Lanzhou General Hospital, Lanzhou, Gansu
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The People's Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University Tumor Hospital of Hebei Province, Shijiazhuang, Hebei
  - Harbin medical university affiliated tumor hospita, Harbin, Heilongjiang
  - Henan Province Tumor Hospital, Luoyan, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The Third Xiangya Hospital Central South University, Changsha, Hunan
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - The General Hospital of Nanhua University, Hengyang, Hunan
  - The First People's Hospital of Changzhou, Changzhou, Jiangsu
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Nantong Cancer Hospital, Nantong, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - Liaoning Province Tumor Hospital, Shenyang, Liaoning
  - Shandong Tumor Hospital, Jinan, Shandong
  - Linyi City Tumor Hospita, Linyi, Shandong
  - Fudan University Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Cancer Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The fourth Military Medical University, Xian, Shanxi
  - Tianjin Medical University Cancer Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Yunnan Province Tumor Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital School of Medical,Zhejiang University, Hangzhou, Zhejiang